CLINICAL TRIAL: NCT02270177
Title: Patients' Satisfaction With Telemedicine Versus Traditional Specialist Consultation for Headache. An Open-labeled Randomized Non-inferiority Study Among Patients With Headache Referred to a Neurologic Outpatient Clinic
Brief Title: Telemedicine Versus Traditional Specialist Consultation for Headache: a Non-inferiority Trial
Acronym: VHS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Collaborators: University of Tromso (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2009/1430 REK sør-øst; FAS nr: 692 (Registry Identifier: Clinical research administrative system (FAS, UNN)); HST959-10 (Registry Identifier: Helse Nord, e-report)
Record Dates: First submitted 2014-10-02; First posted 2014-10-21 (Estimated); Last update posted 2016-06-14 (Estimated); Status verified 2016-05

CONDITIONS: Headaches
Keywords: Headache; Telemedicine; Videoconsultation; Headache-referrals
MeSH Terms: conditions — Headache | interventions — Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Regular consultation (No Intervention): Regular headache consultations
- Videoconsultation (Other): Headache consultations through telemedicine technology
  Interventions: Other: Telemedicine, videoconsultation

INTERVENTIONS:
Other: Telemedicine, videoconsultation — We are investigating the use of videoconsultations (through telemedicine technology) in patients with primary headaches.
  Arms: Videoconsultation

SUMMARY:
Headache is a frequent cause of visits to the GPs office, and the investigators have previously shown that this group accounts for about 20 % of patients referred to a general neurologic outpatient clinic.

To our knowledge, no previous study has investigated whether headache consultation through telemedicine provides equal health care outcomes compared to regular visit to the neurologist. If that's the case, a modern interactive health care system may give simpler and cheaper services for patients, saving travelling costs and community expenses. It may possibly also lead to reduced waiting lists, earlier diagnosis and treatment.

This is an open-labeled randomized non-inferiority trial of headache patients referred to a neurologic clinic in North-Norway. The aim of this study is to determine whether video consultations are non-inferior to regular consultations in diagnosing and treating primary headaches. The null hypothesis is that there is no difference in patient satisfaction between the two groups. The outcome is assessed 3 and 12 months after the neurologic consultation.

Participants will be allocated to either a telemedicine consultation or a regular consultation at the neurologic outpatient clinic in the University Hospital of North-Norway, Tromsø. Both groups will undergo a structured and detailed interview to clarify the diagnosis and establish appropriate treatment. To ensure the best possible representation in the population, our goal is to include at least 70% of all the referred patients that meet the criteria for participation. The randomizations are made through a centralized 8-16 phone line to the research-department in Tromsø, at the University Hospital of North-Norway.

Both primary and secondary endpoints will be assessed in questionnaires sent three and 12 months after the consultation. In addition, the quality of the physicians' referrals and calculations of cost savings by using telemedicine will be evaluated.

The patients' informed consent will always be obtained before data collection. Patients are able to withdraw from the study at any time. Withdrawal will not affect the treatment or follow up. Local research ethics committee (REC) has approved the study.

DETAILED DESCRIPTION:
Epidemiological research shows that over half of Europe's population suffers from headache. Approximately 11% of the population suffers from migraine, over half of the population have tension-type headache, and 4% have chronic daily headaches. There is clear evidence that headaches, and especially migraines, are under- or misdiagnosed. Headache is a frequent cause of visits to the GPs office, and we have previously shown that this group accounts for about 20 % of patients referred to a general neurologic outpatient clinic.

To our knowledge, no previous studies have investigated whether headache consultations through telemedicine provides equal health care outcomes compared to regular visits to the neurologist. If that's the case, a modern interactive health care system may give simpler and cheaper services for patients, saving traveling costs and community expenses. It may possibly also lead to reduced waiting lists, earlier diagnosis and treatment.

This is an open-label randomized non-inferiority study of headache patients referred to our neurologic outpatient clinic. The aim of this study is to determine if video consultations are non-inferior to regular consultations in diagnosing and treating primary headaches. The null hypothesis is that there is no difference in patient satisfaction between the two groups. The outcome is assessed 3 and 12 months after the neurologic consultation. We will allocate participants to either a telemedicine consultation or a regular consultation at the neurologic outpatient clinic in the University Hospital of North-Norway, Tromsø. Both groups will undergo a structured and detailed interview to clarify the diagnosis and establish appropriate treatment. All diagnoses are given by the most up to date version of The International Classification of Headache Disorders (ICHD). We will strive continuously to include all patients who meet the inclusion and exclusion criteria. To ensure the best possible representation in the population, our goal is to include at least 70% of all the referred patients that meet the criteria for participation in this study. The randomizations are made through a centralized 8-16 phone line to the research-department in Tromsø, at the University Hospital of North-Norway.

We will gather the primary and secondary endpoints from the recruited participants by questionnaires sent three and 12 months after the consultation. In addition, we are going to investigate the quality of the physicians' referrals, peoples' use of medications, alternative therapies as well as calculations of cost savings by using telemedicine.

The patients' informed consent will always be obtained before data collection. Patients are able to withdraw from the study at any time. Withdrawal will not affect the treatment or follow up. Local research ethics committee (REC) has approved the study.

ELIGIBILITY:
Inclusion Criteria:

* Females and males ≥16 and ≤65 years of age
* Referred to a neurologist for headache
* No red flags (defined) suggestive of a secondary cause? No known underlying causes of headaches (secondary headaches) according to established criteria
* Referred for diagnostic clarification and / or treatment
* Waiting time ≤ 4 months from the date of the referral
* speaking Norwegian language

Exclusion Criteria:

* Age <16 years or > 65 years of age
* Known underlying cause of the headache or the presence of red flags suggestive of secondary headaches.
* Examined by a neurologist for headaches in a period of 2 years before referral
* Waited longer than 4 months from the date of referral
* Non-Norwegian speaker

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 402 (Actual)
Dates: Start 2012-09; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Number of satisfied participants | change from baseline at 3 months and 12 months
  Are you satisfied with the consultation? Yes/No

SECONDARY OUTCOMES:
VAS satisfaction rating scale | 12 months
  Visual analog satisfaction scale 0-10, where 0 = least satisfied and 10 = most satisfied
VAS pain scale | changes from baseline in VAS at 3 months and 12 months
  Headache measured by a visual analog scale 0-10, 0= no pain, 10=worst pain
HIT-6 | Changes from baseline in HIT 6 at 3 months and 12 months
  Headache impact test
Job situation/occupation | changes from baseline in job situation at 3 months and 12 months
  Job situation/occupation
numbers of consultations during follow up | numbers of consultations from baseline and after 12 months
  numbers of GP-consultations, hospital consultations and admissions
number of pain killers, triptans and other medications for headache | at baseline, after 3 months and after 12 months
  number of medications for headache
headache diagnosis | at baseline, after 3 months and 12 months
  Headache diagnosis after IHS criteria

OTHER OUTCOMES:
Estimation of travelling distances to the neurologic outpatient clinic | travelling distance in kilometers for the neurologic consultation (telemedicine versus regular consultation) and the average travelling distance to the GP during the consecutive 11 months
  travelling distances in kilometers
Expenses saved by using telemedicine | Expenses (travelling, lost income and days absent from work) for the neurologic consultation and the average expenses for GP-consultations during the consecutive 11 months
  Evaluation of the expenses associated with telemedicine compared to regular consultations (travelling expensis, lost earnings, days away from work,
Number of headache days and headaches | change in number of headaches from baseline, at 3 months and 12 months
  Change in number of headache days per month and number of headahces per month
Change in headache feature | Change in headache features from baseline, after 3 months and 12 months
  Is the headahce bether, worse or the same. Is the headahce more intens, less intens or unchanged.

CONTACTS AND LOCATIONS:
Overall Officials: Svein I Bekkelund, MD, PHD, Principal Investigator — Neurologic department, University Hospital of North-Norway, Tromsø and University of Tromsø, Norway
Locations (1):
- Department of Neurology, University Hospital of North Norway, Tromsø, Troms, Norway

REFERENCES:
- [Background] Stovner LJ, Andree C. Prevalence of headache in Europe: a review for the Eurolight project. J Headache Pain. 2010 Aug;11(4):289-99. doi: 10.1007/s10194-010-0217-0. Epub 2010 May 16. PMID 20473702
- [Background] Stovner LJ, Zwart JA, Hagen K, Terwindt GM, Pascual J. Epidemiology of headache in Europe. Eur J Neurol. 2006 Apr;13(4):333-45. doi: 10.1111/j.1468-1331.2006.01184.x. PMID 16643310
- [Background] Stovner LJ, Andree C; Eurolight Steering Committee. Impact of headache in Europe: a review for the Eurolight project. J Headache Pain. 2008 Jun;9(3):139-46. doi: 10.1007/s10194-008-0038-6. Epub 2008 Apr 17. PMID 18418547
- [Background] Bekkelund SI, Albretsen C. Evaluation of referrals from general practice to a neurological department. Fam Pract. 2002 Jun;19(3):297-9. doi: 10.1093/fampra/19.3.297. PMID 11978723
- [Background] Bekkelund SI, Salvesen R. Patient satisfaction with a neurological specialist consultation for headache. Scand J Prim Health Care. 2002 Sep;20(3):157-60. doi: 10.1080/028134302760234609. PMID 12389752
- [Background] Bekkelund SI, Salvesen R. Is uncertain diagnosis a more frequent reason for referring migraine patients to neurologist than other headache syndromes? Eur J Neurol. 2006 Dec;13(12):1370-3. doi: 10.1111/j.1468-1331.2006.01523.x. PMID 17116222
- [Background] Salvesen R, Bekkelund SI. Aspects of referral care for headache associated with improvement. Headache. 2003 Jul-Aug;43(7):779-83. doi: 10.1046/j.1526-4610.2003.03136.x. PMID 12890133
- [Background] Bekkelund SI, Salvesen R; North Norway Headache Study (NNHS). Are headache patients who initiate their referral to a neurologist satisfied with the consultation? A population study of 927 patients--the North Norway Headache Study (NNHS). Fam Pract. 2001 Oct;18(5):524-7. doi: 10.1093/fampra/18.5.524. PMID 11604376
- [Background] Cottrell C, Drew J, Gibson J, Holroyd K, O'Donnell F. Feasibility assessment of telephone-administered behavioral treatment for adolescent migraine. Headache. 2007 Oct;47(9):1293-302. doi: 10.1111/j.1526-4610.2007.00804.x. PMID 17927645
- [Background] Pryse-Phillips W. Evaluating migraine disability: the headache impact test instrument in context. Can J Neurol Sci. 2002 Jun;29 Suppl 2:S11-5. doi: 10.1017/s0317167100001888. PMID 12139080
- [Background] Headache Classification Subcommittee of the International Headache Society. The International Classification of Headache Disorders: 2nd edition. Cephalalgia. 2004;24 Suppl 1:9-160. doi: 10.1111/j.1468-2982.2003.00824.x. No abstract available. PMID 14979299
- [Derived] Bekkelund SI, Muller KI. One-Year Remission Rate of Chronic Headache Comparing Video and Face-to-Face Consultations by Neurologist: Randomized Controlled Trial. J Med Internet Res. 2021 Dec 13;23(12):e30151. doi: 10.2196/30151. PMID 34898455
- [Derived] Muller KI, Alstadhaug KB, Bekkelund SI. A randomized trial of telemedicine efficacy and safety for nonacute headaches. Neurology. 2017 Jul 11;89(2):153-162. doi: 10.1212/WNL.0000000000004085. Epub 2017 Jun 14. PMID 28615434
- [Derived] Muller KI, Alstadhaug KB, Bekkelund SI. Telemedicine in the management of non-acute headaches: A prospective, open-labelled non-inferiority, randomised clinical trial. Cephalalgia. 2017 Aug;37(9):855-863. doi: 10.1177/0333102416654885. Epub 2016 Jun 14. PMID 27301460
- [Derived] Muller KI, Alstadhaug KB, Bekkelund SI. Acceptability, Feasibility, and Cost of Telemedicine for Nonacute Headaches: A Randomized Study Comparing Video and Traditional Consultations. J Med Internet Res. 2016 May 30;18(5):e140. doi: 10.2196/jmir.5221. PMID 27241876